CLINICAL TRIAL: NCT01199107
Title: Maximizing Treatment Outcome and Examining Sleep in Post-traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Southern Methodist University (Other)
Responsible Party: Principal Investigator, Jasper Smits, Ph.D., Principal Investigator, Southern Methodist University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KS10-106
Record Dates: First submitted 2010-09-08; First posted 2010-09-10 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: PTSD; Anxiety; Behavior Therapy; Prolonged Exposure; Exercise; Wellness; Posttraumatic; Stress
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Prolonged Exposure + Exercise (Experimental)
  Interventions: Behavioral: Prolonged Exposure; Behavioral: Exercise
- Prolonged Exposure + Wellness Intervention (Active Comparator)
  Interventions: Behavioral: Prolonged Exposure; Behavioral: Wellness Intervention

INTERVENTIONS:
Behavioral: Prolonged Exposure — 75-90 minute weekly psychotherapy sessions x 12 weeks, focused on gradually confronting distressing trauma-related memories and reminders
Behavioral: Exercise — 30 minutes of moderate-intensity treadmill exercise prior to the Prolonged Exposure
  Arms: Prolonged Exposure + Exercise
Behavioral: Wellness Intervention — 30 minutes of wellness education prior to Prolonged Exposure
  Arms: Prolonged Exposure + Wellness Intervention

SUMMARY:
The purpose of this study is to examine the efficacy of exercise in comparison to wellness education to determine if they can improve the effects of prolonged exposure therapy (PE) in reducing symptoms of anxiety associated with Post-traumatic Stress Disorder (PTSD). In addition, the two strategies (i.e., exercise and wellness education) will be compared in terms of improvements in sleep as well as levels of brain-derived neurotrophic factor (BDNF). BDNF is a protein that helps to support the survival of existing neurons and stimulate the growth new neurons and synapses. BDNF is important to learning and memory in general and therefore may be associated with the learning and memory as it relates to PE and corresponding symptom PTSD improvement.

ELIGIBILITY:
Inclusion Criteria:

* You have PTSD
* You are between the age of 18 and 54 if female or between ages 18 and 44 if male.
* You have written physician approval/medical clearance to participate in an exercise protocol.
* Are currently taking no psychotropic medications or are able and willing to discontinue these medications prior to the first PE session.

Exclusion Criteria:

* You are currently participating in a structured exercise program
* You have severe depression
* You have any history of bipolar disorder, psychotic disorder, or obsessive compulsive disorder;
* You have a diagnosis of eating disorder, or substance abuse or dependence (excluding nicotine) within the past six months
* You have any history of a suicide attempt, or are at significant risk of self-harm or harm to others
* You have ever been diagnosed with organic brain syndrome, mental retardation, or other cognitive dysfunction

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2010-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
PTSD Symptoms | 3 months
  Self-report measure that assesses PTSD Symptoms. Will be assessed at each visit throughout the 3 month protocol.

SECONDARY OUTCOMES:
Sleep Quality | 3 months
  Sleep measure that will be assessed twice (at the beginning and end of the 3 month protocol).
BDNF (by blood sample) | 3 months
  Small blood sample taken twice (at the beginning and end of the 3 month protocol).
General Mood and Anxiety Symptoms | 3 months
  Self-report measure that assesses mood and anxiety. Will be assessed at each visit throughout the 3 month protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- Southern Methodist University, Dallas, Texas, United States

REFERENCES:
- [Derived] Powers MB, Medina JL, Burns S, Kauffman BY, Monfils M, Asmundson GJ, Diamond A, McIntyre C, Smits JA. Exercise Augmentation of Exposure Therapy for PTSD: Rationale and Pilot Efficacy Data. Cogn Behav Ther. 2015;44(4):314-27. doi: 10.1080/16506073.2015.1012740. Epub 2015 Feb 23. PMID 25706090